CLINICAL TRIAL: NCT05490862
Title: Inflammatory Status of Monocytes in Obesity: Association With Atherosclerosis Indicators and the Effectiveness of Weight Loss
Brief Title: Inflammatory Status of Monocytes in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Yurgita R. Varaeva, MD, MRes, Dr, Research Fellow, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-25-00414
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: obesity; Cardiovascular risk factors; atherosclerosis; Inflammation; Monocytes; Cytokines
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Atherosclerosis; Inflammation

STUDY DESIGN:
Intervention Model Description: Match pairs Parallel group Double-control design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obese Weight Loss group (Experimental): Low-calorie diet and regular physical trainings will be administered to obese participants (BMI >30kg/m^2).
  Interventions: Behavioral: Lifestyle Modification
- Obese Control group (Active Comparator): Traditional weight loss recommendations will be provided to obese participants (BMI >30kg/m^2)
  Interventions: Behavioral: Traditional Recommendations
- Lean Control group (No Intervention): The data of these subjects will be used as a control

INTERVENTIONS:
Behavioral: Lifestyle Modification — An individualized low-calorie diet is characterized by sugars and starchy food intake restriction, 500 kcal daily energy deficit for 12 weeks (3 months).
  Regular physical activity is represented by individualized 30 minutes trainings on an anti-gravity treadmill 3 workouts per week for 12 weeks with individual targets of stepping activity, which will be evaluated according to personal fitness monitoring data
  Arms: Obese Weight Loss group
Behavioral: Traditional Recommendations — The list of traditional diet and physical activity recommendations for patients with obesity
  Arms: Obese Control group

SUMMARY:
The study of the pro-inflammatory activation of circulating monocytes/macrophages in obesity is the main problem of this project. The investigation of pro-inflammatory activation of monocytes and determination of the level of mitochondrial genome mutations, assessment of traditional CVD risk factors and the degree of cardiovascular risk and atherosclerosis indicators and their association will be investigated in dynamics on 12-weeks weight loss.

DETAILED DESCRIPTION:
Obesity is one of the main risk factors for cardiovascular disease (CVD), which occupy the first place in the overall structure of mortality in developed countries, and therefore it is a serious medical and social problem and an urgent research topic in modern science. Inflammation is one of the key factors in the development of cardiovascular complications of obesity, in particular atherogenesis. Currently, the mechanisms of inflammation in obesity are widely studied, in experimental studies, special attention is paid to the study of macrophages of adipose tissue, their inflammatory activation and their role in the development of obesity-associated pathological conditions. Circulating monocytes in dense tissue differentiate into macrophages and play an important role in the pathogenesis of chronic inflammation. Increased pro-inflammatory activation of macrophages in the focus of inflammation can cause chronic inflammation and contribute to the development of atherosclerotic lesions in the vascular wall. Mitochondrial dysfunction may play a special role in the proinflammatory activation of monocytes since it leads to the accumulation of oxygen radicals and activates the excessive secretion of inflammatory mediators. Mitochondrial genome mutations are one of the possible mechanisms leading to the development of mitochondrial dysfunction. Previously, atherosclerosis-associated mutations of the mitochondrial genome were identified, however, in obesity, the level of mitochondrial heteroplasmy has not been studied. Weight loss is associated with a decrease in cardiovascular risk; however, the mechanisms of the cardioprotective effects of weight loss are not fully understood. The anti-inflammatory effects of vigorous exercise in obesity are being actively studied. The study of the pro-inflammatory activation of circulating monocytes/macrophages in obesity is the main problem of this project. The following tasks will be solved within the framework of the project: 1. Investigation of pro-inflammatory activation of monocytes and determination of the level of mitochondrial genome mutations in obese individuals. 2. Comprehensive assessment of the association of monocyte activation, mitochondrial genome mutations and traditional CVD risk factors and the degree of cardiovascular risk and atherosclerosis indicators in obese individuals. 3. Study on the effect of weight loss after a 3-month course of body weight loss, consisting of a set of physical exercises in combination with a low-calorie diet on the inflammatory status of monocytes in obese individuals.

As a result of the project, data on the inflammatory status of monocytes in obesity will be obtained and published, the effect of pro-inflammatory activation of monocytes, mitochondrial genome mutations in combination with traditional CVD risk factors on indicators of atherosclerosis and cardiovascular risk in obese individuals will be investigated. Data on the effect of a weight loss intervention (a combination of exercise complex and low-calorie diet) on the inflammatory status of monocytes will be obtained and published. The study of cellular markers of inflammation and the identification of mitochondrial genome mutations in obese individuals will deepen the understanding of the mechanisms of chronic inflammation in obesity and obesity-associated cardiovascular complications. The study of the effect of weight loss on the inflammatory status of monocytes - key cells in the development of chronic inflammation - may become a promising direction for the development of approaches for personalized pathogenetic therapy of obesity and prevention of obesity-associated cardiovascular complications.

ELIGIBILITY:
Obese Weight Loss and Control groups Inclusion Criteria:

• BMI ≥30 kg/m2

Lean Control group Inclusion Criteria:

• BMI <25 kg/m2

Exclusion Criteria:

* Diabetes Mellitus
* Cancer
* Uncontrolled Hypertension
* Decompensated liver or kidney disease
* III-IV classes of Chronic Heart Failure
* Other chronic diseases (except CVDs) on permanent treatment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Changes of pro-inflammatory macrophages activation | Twice: Baseline, treatment week 12
  The measurement of basal and lipopolysaccharide-induced tumor necrosis factor-α and interleukin-1β levels in the culture of cluster differentiation 14+ cells obtained from participants blood samples
Mitochondrial genome mutations | One time measurement (baseline)
  The assessment of mtDNA mutation heteroplasmy m.652delG, m.1555A>G, m.3336T>C, m.3256C>T, m.5178C>A, m.12315G>A, m.13513G>A, m.14459G>A , m.14846G>A и m.15059G>A by real-time polymerase chain reaction

SECONDARY OUTCOMES:
Changes of body mass | Twice: Baseline, treatment week 12
  Includes repeated assessment of body mass (kg) and calculation of percentage of weight loss.
Changes of body fat mass | Twice: Baseline, treatment week 12
  Includes repeated assessment of body fat mass (%) by bio-impedancemetry body composition analysis and calculation of fat mass loss.
Changes of skeletal muscle mass | Twice: Baseline, treatment week 12
  Includes repeated assessment of skeletal muscle mass (%) by bio-impedancemetry body composition analysis and calculation of muscle mass changes (positivo or negative).
Changes of Serum Cholesterol levels | Twice: Baseline, treatment week 12
  The measurement of serum total cholesterol and cholesterol sbgroups levels by standard laboratory procedures. The decrease of cholesterol levels is considereed as positeve effect.
Framingham Risk Score | Twice: Baseline, treatment week 12
  The assessment of estimated 10-year cardiovascular risk (%) according to the Framingham Risk Score that varies from less than 10% (low risk) to more than 20% (high risk). The reduction od risk will be considered as positive effect of intervention.
Intima-media thickness | One time measurement (baseline)
  The assessment of intima-media thickness of common carotid artery evaluated by B-mode ultrasound imagining.

CONTACTS AND LOCATIONS:
Overall Officials: Yurgita R Varaeva, MD, MRes, Principal Investigator — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Locations (1):
- Department of Cardiovascular Pathology and Diet, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Per reasonable request to principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after study completion
Access Criteria: Per reasonable request
URL: http://www.ion.ru